CLINICAL TRIAL: NCT02971995
Title: Trimodal (18)F-choline-PET/mpMRI/TRUS Targeted Prostate Biopsies in Prostate Cancer Patients
Brief Title: Trimodal (18)F-choline-PET/mpMRI/TRUS Targeted Prostate Biopsies
Acronym: PROSTEPIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OBS025
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2015-06

CONDITIONS: Prostatic Neoplasm; Positron-Emission Tomography; Fluorocholine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostate cancer/TEP scan (Experimental)
  Interventions: Device: PET Scan ou TEP-TDM
- Prostate cancer/mpMRI (Active Comparator)
  Interventions: Device: mpMRI

INTERVENTIONS:
Device: PET Scan ou TEP-TDM — Performance of the PET/CT using Flurocholine in order to detect the localization of the pathological fixation of the tracer and to determine the place where to take the biopsy
  Arms: Prostate cancer/TEP scan
Device: mpMRI — Performance of the mpMRI in order to determine the place where to take the biopsy
  Arms: Prostate cancer/mpMRI

SUMMARY:
Prostate cancer is the first cancer in humans (25%). The most widely used tracer in oncology, the 18-Fluoro DeoxyGlucose does not allow the study of prostatic neoplasia. On the other hand, Choline, which is an amino alcohol, is involved in the synthesis of cell membranes and has an affinity for prostate cells. Its concentration is directly proportional to cell proliferation. The analogue of choline has the advantage of having a rapid and stable accumulation over time in cancer cells, with a rapid urinary excretion (4 minutes after injection).

The goal of this study is to assess the feasibility and the accuracy for targeting image guided prostate biopsy to detect prostate cancer after Imaging fusion of choline-PET/CT compared to 1.5T multiparametric magnetic resonance imaging (mpMRI) with 3D-transrectal ultrasound (TRUS) .

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of prostate cancer
* Patients who performed prostate mpMRI and F-Choline 18 PET scan
* Patient capable of receiving clear informations
* Patient giving a written consent for their participation via a consent signed by both parents of the patient (or legal tutor)
* Patient covered by a healthcare insurance

Exclusion Criteria:

* Patients without suspect image of neoplasia after mpMRI and F-Choline 18 PET scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of image guided prostate biopsy in the zones detected by the TEP scan | at inclusion

SECONDARY OUTCOMES:
Number of image guided prostate biopsy in the zones detected by the mpMRI | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Bonnal, MD, Principal Investigator — GHICL

IPD SHARING:
Plan to Share IPD: No